CLINICAL TRIAL: NCT02813980
Title: Neural Circulatory and Respiratory Control in Patients With Epilepsy and the Risk of Sudden Unexpected Death.
Brief Title: Neural Circulatory Control and SUDEP Risk.
Acronym: NC-SUDEP
Status: Active, not recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Virend Somers, MD, PhD, PI, Mayo Clinic
Other Study IDs: 15-001421
Record Dates: First submitted 2016-06-22; First posted 2016-06-27 (Estimated); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Epilepsy; Seizures
Keywords: SUDEP; Sudden cardiac death; Sudden unexpected death in epilepsy; Sleep; Polysomnography; Autonomic; Cardiovascular
MeSH Terms: conditions — Epilepsy; Seizures; Sudden Unexpected Death in Epilepsy; Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and plasma to be stored for future biomarker based studies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High SUDEP-7 score: Patients with epilepsy who have a high SUDEP-7 score
- Low SUDEP-7 score: Patients with epilepsy who have a low SUDEP-7 score

SUMMARY:
The investigators believe epilepsy alters the way the body controls blood pressure, heart rate and breathing, and these changes increase the risk of sudden unexpected death in patients with epilepsy (SUDEP). SUDEP-7 is a risk scoring tool which may correlate with these changes to the heart and blood vessels. This research study measures those differences which may help identify new markers to help predict those patients at greatest risk in the future.

DETAILED DESCRIPTION:
The investigators overall goals are to determine whether measures of neural-circulatory control during the interictal waking and sleep states, as well as during the ictal/peri-ictal periods, are associated with SUDEP-7 score risk profiles in refractory epilepsy patients, and to translate these measures into tools for risk-stratification and preventative strategies for SUDEP.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-90
* Able to consent

Exclusion Criteria:

* History of non-epileptic spells/seizures,
* Children/adolescents under age 18 years
* Pregnancy
* Non-compliance with Epilepsy Monitoring Unit safety procedures
* Unable to consent
* History of dysautonomia
* Chronic Obstructive Pulmonary Disease (COPD)
* Asthma (active requiring therapy)
* Pulmonary hypertension
* Known Structural Heart Disease
* Heart failure
* Myocardial infarction
* Stroke
* Seizures due to traumatic injury
* Prior surgery for epilepsy
* Vasculitis
* Raynaud's
* Smoking (current or within the last 6 months)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with epilepsy.
Sampling Method: Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Abnormal neural circulatory control in patients with epilepsy and high SUDEP-7 scores compared to patients with epilepsy and low SUDEP-7 scores. | 24 hours
Abnormal neural and respiratory control in the ictal and peri-ictal phase of patients with epilepsy and a high SUDEP-7 score when compared to patients with epilepsy and a low SUDEP-7 score. | 3-7 days

CONTACTS AND LOCATIONS:
Overall Officials: Virend K Somers, MD PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials